CLINICAL TRIAL: NCT06775977
Title: Ultrasound Contrast-Enhanced Accurate Diagnosis of Preoperative Staging of Bladder Cancer: a Prospective, Observational Study
Brief Title: Ultrasound Contrast-Enhanced Accurate Diagnosis of Preoperative Staging of Bladder Cancer
Acronym: UCEADP-BCS
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qiyun Ou, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-145-01; Grant No.2023CSM003 (Other Grant/Funding Number: the Guangdong Yiyang Healthcare Charity Foundation)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer; Staging; Contrast Enhanced Ultrasound
Keywords: Bladder Cancer; Contrast-Enhanced Ultrasonography
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Contrast-enhanced Ultrasonography: To evaluate the diagnostic accuracy of CEUS for the preoperative staging of bladder cancer, which would benefit the implementation of efficient therapeutic strategies.
  Interventions: Diagnostic Test: Contrast Enhanced Ultrasound (CEUS)

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Ultrasound (CEUS) — Contrast Enhanced Ultrasound (CEUS) refers to the observation under ultrasound after the injection of ultrasound contrast agents, such as SonoVue or Lumason.

SUMMARY:
Ultrasound and magnetic resonance imaging (MRI) technologies have become essential tools for the diagnosis and preoperative staging assessment of bladder cancer. However, establishing a precise system suitable for clinical application remains a significant challenge, and accurate prediction of bladder cancer staging is not yet possible. Therefore, exploring a system for the precise diagnosis of preoperative staging of bladder cancer using ultrasound contrast enhancement or a combination of ultrasound contrast enhancement and MRI is of great importance. The applicant has previously demonstrated the accuracy of multimodal data analysis in the diagnosis and prediction of malignant tumors. Preliminary results from this study have shown that ultrasound contrast enhancement has a high diagnostic efficacy for the preoperative staging assessment of bladder cancer, with a high area under the curve (AUC) of 0.88, sensitivity of 83.3%, specificity of 92.5%, and accuracy of 90.8%. In this project, the applicant intends to further expand the sample size and, based on the combination of ultrasound contrast enhancement and MRI, develop a precise diagnostic system for the preoperative staging of bladder cancer to aid clinical treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* (a) eligible patients should be 18-year-old or older;
* (b) patients should have a histologically or cytologically confirmed diagnosis of primary bladder cancer;
* (c) patients should not have had any surgery, chemotherapy, immunotherapy, or any therapy before CEUS diagnosis.

Exclusion Criteria:

* (a) participants with confirmed to have no carcinoma of the bladder;
* (b) participants with previous pelvic surgery, who had undergone therapy, any bladder surgery, or had received chemotherapy, radiotherapy or immunotherapy;
* (c) participants diagnosed with tumor recurrence or metastasis; (d) participants who were allergic to ultrasound contrast agents or could not tolerate CEUS examination, for instance, with recent myocardial infarction, angina pectoris, cardiac insufficiency, severe cardiac arrhythmia, a right/left cardiac shunt, severe pulmonary hypertension, uncontrolled systemic hypertension, acute respiratory distress syndrome, or chronic obstructive pulmonary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have a histologically or cytologically confirmed diagnosis of primary bladder cancer
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Muscle Invasion in Bladder Cancer | within 3 minutes
  To evaluate the preoperative staging of bladder cancer，whether it is non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancers (MIBC)

CONTACTS AND LOCATIONS:
Overall Officials: Luo, Prof., Study Director — Department of Ultrasound in Medicine, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, Analytic Code